CLINICAL TRIAL: NCT05855317
Title: Association Between the Level of Extracellular Vesicle - Associated Tissue Factor and the Occurence of Pulmonary Embolism in Patients With Acute Respiratory Distress Syndrome
Brief Title: Association Between the Level of EV-TF and the Occurence of Pulmonary Embolism in Patients With ARDS
Acronym: THROMBO-EVTF
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM22_0440; ID-RCB (Other: 2023-A00413-42)
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pulmonary embolism: The presence of pulmonary embolism is determined from a CT scan realized between Day 5 and Day 28.
  Interventions: Other: Blood sample
- Patients without pulmonary embolism: The absence of pulmonary embolism is determined from a CT scan realized between Day 5 and Day 28.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Additional blood samples will be taken on a catheter, used for standard care.

SUMMARY:
In this study, 120 patients with Acute Respiratory Distress Syndrome (ARDS) will be included on a two years-period in an intensive care unit (Assistance Publique des Hôpitaux de Marseille, France). Those patients will benefit from a blood test at inclusion in order to measure several coagulation biomarkers, including EV-TF. Subsequently, these patients will be treated according to the usual practices of the department, following recommendations. Patients who received an injected CT scan between Day 5 and Day 28 will be divided into two groups based on the presence or absence of a pulmonary embolism on imaging. The measured values of EV-TF levels and other studied biomarkers will be compared between these two groups in order to detect a possible association between them and the diagnosis of pulmonary embolism. It should be noted that patients receiving an injected CT-scan between Day 5 and Day 7 will be included in the main analysis while those receiving it between Day 8 and Day 28 will be included in the secondary analysis. Others will be excluded from any analysis. At the same time, several collections of clinical data will be carried out: on Day 1, Day 7, Day 28, and on the day of the CT scan if it is performed at another time.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older,
* Patient who has given his/her non-opposition to participate in this study, or alternatively, patient for whom a relative has given his/her non-opposition to participate in this study,
* Patient admitted to intensive care for less than 24 hours,
* Patient with ARDS according to the Berlin criteria,

  * Hypoxemia with PaO2/FiO2 ratio ≤ 300 on mechanical ventilation under PEEP ≥ 5 cmH2O,
  * Bilateral alveolar-interstitial opacities on chest imaging (chest X-ray or CT),
  * Exclusion of a cardiogenic cause on echocardiography,
  * Acute or subacute onset within 7 days based on the clinical-radiological profile.

Exclusion Criteria:

* Positive SARS-CoV-2 PCR in a pharyngeal or respiratory sample (cytobacteriological examination of sputum, bronchial aspiration or bronchoalveolar lavage) prior to admission to the intensive care unit,
* Patient with a pathology affecting the coagulation process or endothelial function (hemophilia, von Willebrand disease, etc.),
* Patient receiving curative anticoagulant treatment before admission to the intensive care unit,
* Patient undergoing extracorporeal veno-venous respiratory assistance (ECMO-VV) before admission to the intensive care unit,
* Patient undergoing extra-renal purification with systemic anticoagulation with heparin before admission to the intensive care unit,
* Persons referred to in articles L. 1121-5 to L. 1121-8 of the Public Health Code (minor patients, adult patients under tutorship or guardianship, patients deprived of their liberty, pregnant or nursing women),
* Moribund patients for whom the life expectancy is less than 24 hours according to the opinion of the investigating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS admitted to the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Difference in EV-TF levels at inclusion between patients with and without pulmonary embolism at day 7 postinclusion | Day 7
  EV-TF level is determined from a blood sample realized at inclusion and the presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.

SECONDARY OUTCOMES:
Difference in EV-TF levels at inclusion between patients with and without pulmonary embolism at day 28 postinclusion | Day 28
  EV-TF level is determined from a blood sample realized at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Difference in EV-TF levels at inclusion between patients with and without venous thrombo-embolic disease at day 7 postinclusion | Day 7
  EV-TF level is determined from a blood sample realized at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Difference in EV-TF levels at inclusion between patients with and without venous thrombo-embolic disease at day 28 postinclusion | Day 28
  EV-TF level is determined from a blood sample realized at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Association between EV-TF levels and patient prognosis | Day 60
  EV-TF level is determined from a blood sample realized at inclusion. Patient prognosis is based on the duration of intensive care unit stay, on the duration of hospital stay, and on death.
Association between EV-TF level and alveolar dead space at inclusion | Day 1
  EV-TF level is determined from a blood sample realized at inclusion. Alveolar dead space is obtained by volumetric capnography at inclusion.
Association between EV-TF level and alveolar dead space at day 7 postinclusion | Day 7
  EV-TF level is determined from a blood sample realized at inclusion. Alveolar dead space is obtained by volumetric capnography at day 7 postinclusion.
Association between EV-TF level and alveolar dead space at day 28 postinclusion | Day 28
  EV-TF level is determined from a blood sample realized at inclusion. Alveolar dead space is obtained by volumetric capnography at day 28 postinclusion.
Association between EV-TF level and alveolar dead space at thoracic CT scan day | Between day 5 and day 28
  EV-TF level is determined from a blood sample realized at inclusion. Alveolar dead space is obtained by volumetric capnography at day of CT-scan.
Optimal threshold value of EV-TF associated with the occurrence of pulmonary embolism. | Day 28
  EV-TF level is determined from a blood sample realized at inclusion. Occurrence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Optimal threshold value of EV-TF associated with the occurrence of venous thrombo-embolic disease. | Day 28
  EV-TF level is determined from a blood sample realized at inclusion. Occurrence of venous thrombo-embolic disease pulmonary embolism is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Optimal threshold value of EV-TF associated with the occurrence of death | Day 60
  EV-TF level is determined from a blood sample realized at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of Willebrand antigen at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of ADAMTS13 activity at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of circulating levels of antithrombin (coagulation inhibitor) at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of circulating levels of protein C (coagulation inhibitor) at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of circulating levels of protein S (coagulation inhibitor) at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of D-dimers (circulating fibrinolytic potential) at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of fibrin monomers (circulating fibrinolytic potential) at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of circulating PAI-1 (circulating fibrinolytic potential) at inclusion on the occurrence of pulmonary embolism at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism from a CT scan realized during the first week of patient care in intensive care unit.
Predictive value of Willebrand antigen at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of ADAMTS13 activity at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating levels of antithrombin (coagulation inhibitor) at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating levels of protein C (coagulation inhibitor) at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating levels of protein S (coagulation inhibitor) at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of D-dimers (circulating fibrinolytic potential) at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of fibrin monomers (circulating fibrinolytic potential) at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating PAI-1 (circulating fibrinolytic potential) at inclusion on the occurrence of pulmonary embolism at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of pulmonary embolism is determined from a CT scan realized during the first 28 days of patient care in intensive care unit.
Predictive value of Willebrand antigen at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of ADAMTS13 activity at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of circulating levels of antithrombin (coagulation inhibitor) at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of circulating levels of protein C (coagulation inhibitor) at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of circulating levels protein S (coagulation inhibitor) at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of D-dimers (circulating fibrinolytic potential) at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of fibrin monomers (circulating fibrinolytic potential) at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of circulating PAI-1 (circulating fibrinolytic potential) at inclusion on the occurrence of venous thrombo-embolic disease at day 7. | Day 7
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first week of patient care in intensive care unit.
Predictive value of Willebrand antigen at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of ADAMTS13 activity at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating levels of antithrombin (coagulation inhibitor) at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating levels of protein C (coagulation inhibitor) at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating levels of protein S (coagulation inhibitor) at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of D-dimers (circulating fibrinolytic potential) at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of fibrin monomers (circulating fibrinolytic potential) at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of circulating PAI-1 (circulating fibrinolytic potential) at inclusion on the occurrence of venous thrombo-embolic disease at day 28. | Day 28
  This biomarker is quantified from the blood sample collected at inclusion. The presence of venous thrombo-embolic disease is determined from an echo-doppler realized during the first 28 days of patient care in intensive care unit.
Predictive value of Willebrand antigen at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of ADAMTS13 activity at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of of circulating levels of antithrombin (coagulation inhibitor) at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of of circulating levels of protein C (coagulation inhibitor) at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of of circulating levels of protein S (coagulation inhibitor) at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of D-dimers (circulating fibrinolytic potential) at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of fibrin monomers (circulating fibrinolytic potential) at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).
Predictive value of circulating PAI-1 (circulating fibrinolytic potential) at inclusion on the patients' death. | Day 60
  This biomarker is quantified from the blood sample collected at inclusion. Occurrence of death is measured during the 2 months of follow up (or when the patient is discharged from hospital, if earlier).

CONTACTS AND LOCATIONS:
Overall Officials: François Cremieux, Study Director — AP-HM
Locations (1):
- Service Médecine intensive et réanimation, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided